CLINICAL TRIAL: NCT04708184
Title: A Randomized, Open-label, 3-period, Single-dose, Crossover Study in Healthy Adult Subjects to Assess the Relative Bioavailability of GLPG3970 Given as an Oral Tablet Formulation Versus the Oral Solution Formulation of GLPG3970 and to Assess the Effect of Food on the Oral Tablet Formulation.
Brief Title: A Study to Assess Relative Bioavailability of and Effect of Food on a New Oral Tablet Formulation of GLPG3970
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG3970-CL-104; 2020-003997-34 (EudraCT Number)
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GLPG3970 solution (Experimental): Single oral dose of GLPG3970 in fasted conditions
  Interventions: Drug: GLPG3970 oral solution
- GLPG3970 tablet fasted (Experimental): Single oral dose of GLPG3970 in fasted conditions
  Interventions: Drug: GLPG3970 tablet
- GLPG3970 tablet fed (Experimental): Single oral dose of GLPG3970 in fed conditions
  Interventions: Drug: GLPG3970 tablet

INTERVENTIONS:
Drug: GLPG3970 oral solution — GLPG3970 for oral administration
  Arms: GLPG3970 solution
Drug: GLPG3970 tablet — GLPG3970 for oral administration
  Arms: GLPG3970 tablet fasted; GLPG3970 tablet fed

SUMMARY:
This is a study to assess the relative bioavailability of a GLPG3970 oral tablet formulation compared to an oral solution formulation and the effect of food on the bioavailability of a single dose of the oral tablet formulation of GLPG3970. It will also evaluate the safety and tolerability of a single dose of GLPG3970.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age (extremes included), on the date of signing the informed consent form .
* A body mass index between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to randomization. Total bilirubin, aspartate aminotransferase, and alanine aminotransferase must be no greater than 1.5x upper limit of normal range. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator.

This list only contains the key inclusion criteria.

Exclusion Criteria:

* Known hypersensitivity to investigational product (IP) ingredients or history of a significant allergic reaction to IP ingredients as determined by the investigator.

This list only contains the key exclusion criterion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3970 | Between Day 1 pre-dose and Day 4
  To assess the bioavailability (BA) of a GLPG3970 oral tablet formulation (test) relative to that of an oral solution formulation (reference). To assess the effect of food on BA of a single oral dose of the oral tablet formulation of GLPG3970.
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) | Between Day 1 pre-dose and Day 4
  To assess the BA of a GLPG3970 oral tablet formulation (test) relative to that of an oral solution formulation (reference). To assess the effect of food on BA of a single oral dose of the oral tablet formulation of GLPG3970.
Area under the plasma concentration-time curve from time zero until the last observed quantifiable concentration (AUC0-t) | Between Day 1 pre-dose and Day 4
  To assess the BA of a GLPG3970 oral tablet formulation (test) relative to that of an oral solution formulation (reference). To assess the effect of food on BA of a single oral dose of the oral tablet formulation of GLPG3970.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) by Severity | From Day 1 through study completion, an average of 1 month
  To evaluate the safety and tolerability of a single dose of GLPG3970.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Tankisheva, MD, Study Director — Galapagos NV
Locations (1):
- Biotral Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No